CLINICAL TRIAL: NCT00563446
Title: Conversion From Once Weekly Recombinant Human Erythropoietin to Once Monthly Darbepoetin Alfa for the Treatment of Renal Anemia in Continuous Ambulatory Peritoneal Dialysis Patients
Brief Title: Study of the Efficacy of Darbepoetin Alfa in the Treatment of Renal Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Kirin Pharmaceutical (Asia) CO., LTD (Unknown)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KWC/EX/05-041; HARECCTR0500029
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Anemia; Kidney Failure, Chronic; Peritoneal Dialysis, Continuous Ambulatory
Keywords: Anemia; End-stage renal failure; Continuous ambulatory peritoneal dialysis
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa

SUMMARY:
Anaemia is a common consequence of chronic renal failure. Darbepoetin alfa is a unique erythropoietic protein that stimulates erythropoiesis by the same mechanism as endogenous erythropietin and conventional recombinant human erythropoietin (rHuEPO). Darbepoetin alfa has been shown to have a serum half-life 3-fold longer than that of rHuEPO, which allows dosing at extended intervals and less frequent injection.

The objective is to evaluate the efficacy and safety of darbepoetin alfa therapy given at an extended once monthly dosing interval in the treatment of renal anaemia in continuous ambulatory peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients on continuous ambulatory peritoneal dialysis
* Patients receiving subcutaneous recombinant human erythropoietin (rHuEPO)
* Patients with haemoglobin level ?10 g/dL and remain stable for the past 3 months while receiving rHuEPO

Exclusion Criteria:

* Uncontrolled hypertension
* Severe congestive heart failure (NYHA class III or IV)
* Grand mal epilepsy
* Any kind of blood loss causing Fe depletion
* Presence of infection, either acute or chronic, or inflammatory conditions within 3 months preceding the study
* Malignancy
* Aluminum toxicity
* Severe hyperparathyroidism with marrow fibrosis or osteitis fibrosa _ PTH > 20 times of normal
* Vitamin B12 or folate deficiency _ MCV > 100fL
* Haemolysis
* Marrow dysfunction e.g. aplastic anaemia, myelodysplastic syndrome, multiple myeloma, etc
* Thalassaemia major, intermediate or minor, or red cell enzyme defects
* Blood transfusion within 3 months preceding the study
* Pregnancy or lactating mothers

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2005-07; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | Over 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel KS Fung, Dr, Principal Investigator — Division of Nephrology, Medicine & Geriatrics, Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, Hong Kong, China